CLINICAL TRIAL: NCT02625428
Title: Does Contrast-Enhanced Ultrasound Positively Influence Selection of Biopsy Sites When Evaluating Transplant Kidneys?
Brief Title: IRB 14-009240, Does CEUS Positively Influence Selection of Biopsy Sites When Evaluating Transplant Kidneys?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Scott Kriegshauser, M.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14-009240
Record Dates: First submitted 2015-11-10; First posted 2015-12-09 (Estimated); Results first posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Transplantation, Kidney
MeSH Terms: interventions — FS 069; Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- For Cause (Experimental): For cause biopsies to evaluate a recent rise in serum creatinine.
  Interventions: Drug: Optison; Diagnostic Test: Ultrasound (US); Diagnostic Test: Contrast-enhanced ultrasound (CEUS)
- Surveillance (Experimental): Surveillance biopsies done after transplant mostly looking for subclinical rejection.
  Interventions: Drug: Optison; Diagnostic Test: Ultrasound (US); Diagnostic Test: Contrast-enhanced ultrasound (CEUS)

INTERVENTIONS:
Drug: Optison
  Other Names: ultrasound contrast agent
Diagnostic Test: Ultrasound (US) — A routine diagnostic and color-Doppler US. A Doppler ultrasound is a noninvasive test that can be used to estimate the blood flow through your blood vessels by bouncing high-frequency sound waves (ultrasound) off circulating red blood cells. A regular ultrasound uses sound waves to produce images, but can't show blood flow.
Diagnostic Test: Contrast-enhanced ultrasound (CEUS) — Contrast-enhanced ultrasound (CEUS) is the application of ultrasound contrast medium to traditional medical sonography. Ultrasound contrast agents rely on the different ways in which sound waves are reflected from interfaces between substances. This may be the surface of a small air bubble or a more complex structure.

SUMMARY:
This is a pilot study to investigate whether contrast-enhanced ultrasound (CEUS) may help evaluate segmental differences in renal perfusion better than Doppler Ultrasound and thus help direct the biopsy to the most abnormal part of the renal cortex. This should maximize detection and increase the odds of demonstrating the true grade/severity of the histopathological abnormality.

ELIGIBILITY:
Inclusion

* Ability to provide informed consent
* Male and female >18 years
* Patients undergoing renal transplant ultrasound-guided percutaneous biopsy within 24 months post transplant including patients undergoing biopsy to evaluate a recent rise in serum creatinine so called for cause biopsies and patients undergoing routine protocol (surveillance) biopsies without other evident of renal dysfunction

Exclusion:

* Pregnant women or women who are nursing an infant are not able to participate in this study
* Known patent forearm ovale (PFO)
* Significant heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Kriegshauser, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- For Cause: For cause biopsy to evaluate a recent rise in serum creatinine.
  Optison
  Ultrasound (US): A routine diagnostic and color-Doppler US. A Doppler ultrasound is a noninvasive test that can be used to estimate the blood flow through your blood vessels by bouncing high-frequency sound waves (ultrasound) off circulating red blood cells. A regular ultrasound uses sound waves to produce images, but can't show blood flow.
  Contrast-enhanced ultrasound (CEUS): Contrast-enhanced ultrasound (CEUS) is the application of ultrasound contrast medium to traditional medical sonography. Ultrasound contrast agents rely on the different ways in which sound waves are reflected from interfaces between substances. This may be the surface of a small air bubble or a more complex structure.
- Surveillance: Surveillance biopsy done after transplant mostly looking for subclinical rejection.
  Optison
  Ultrasound (US): A routine diagnostic and color-Doppler US. A Doppler ultrasound is a noninvasive test that can be used to estimate the blood flow through your blood vessels by bouncing high-frequency sound waves (ultrasound) off circulating red blood cells. A regular ultrasound uses sound waves to produce images, but can't show blood flow.
  Contrast-enhanced ultrasound (CEUS): Contrast-enhanced ultrasound (CEUS) is the application of ultrasound contrast medium to traditional medical sonography. Ultrasound contrast agents rely on the different ways in which sound waves are reflected from interfaces between substances. This may be the surface of a small air bubble or a more complex structure.
Period: Overall Study
Arm/Group | For Cause | Surveillance
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | For Cause | Surveillance | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (13.4) | 50.8 (14.1) | 52.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 12 | 16 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 3.3 (1.9) | 1.5 (0.4) | 2.4 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Biopsy
Description: Number of subjects with abnormal biopsies in either the primary or secondary biopsy location, by diagnosis from a clinical pathologist
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | For Cause | Surveillance
Number analyzed (Participants) | 20 | 20
Participants | 10 | 7

2. Secondary Outcome: Number of Patients With a Higher Degree of Renal Transplant Rejection Using Multiple Biopsies Compared to a Single Biopsy.
Time Frame: 1 year
Population: This outcome measure was not evaluated or analyzed as all subjects received multiple biopsies
Arm/Group | For Cause | Surveillance
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of biopsy to 1 week post biopsy.
Arm/Group | For Cause | Surveillance
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | For Cause (N=20) | Surveillance (N=20)
Major Bleeding Complications (Blood and lymphatic system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT02625428/Prot_SAP_000.pdf